CLINICAL TRIAL: NCT05579171
Title: A Single Center, Evaluator-Blinded, Split-Face, Randomized Clinical Trial of Combination Treatment With Fractional Picosecond 755nm Alexandrite Laser and Radiofrequency Microneedling for Atrophic Acne Scars
Brief Title: Lasers to Aid in Treatment of Acne Scars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Collaborators: Cynosure, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Potenza-Picosure-Acne Scars
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Acne Scars
Keywords: Acne; Scars; Acne Scars; Lasers; Cosmetic
MeSH Terms: conditions — Acne Vulgaris; Cicatrix | interventions — Lasers, Solid-State

STUDY DESIGN:
Intervention Model Description: Enrolled subjects will be randomized to receive picosecond 755 nm Alexandrite laser treatment to either the left or right facial half. The subjects will then undergo full face radiofrequency microneedling (RFM).
Who Masked: Care Provider, Investigator
Masking Description: Blinded Investigator will be unaware of which side received both treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Left Side Treatment with picosecond 755nm Alexandrite laser (Experimental): Subjects will have their left side of face treated with picosecond 755nm Alexandrite laser then will undergo full face radiofrequency microneedling.
  Interventions: Device: Picosecond 755nm Alexandrite Laser
- Right Side Treatment with Picosecond 755NM Alexandrite laser (Experimental): Subjects will have their right side of face treated with picosecond 755nm Alexandrite laser then will undergo full face radiofrequency microneedling.
  Interventions: Device: Picosecond 755nm Alexandrite Laser

INTERVENTIONS:
Device: Picosecond 755nm Alexandrite Laser — Fractionated picosecond technology has been shown to lead to statistically significant improvement in atrophic, facial acne scars after 4-6 treatment sessions with minimal pain or downtime
  Other Names: Alex Laser
  Arms: Left Side Treatment with picosecond 755nm Alexandrite laser
Device: Picosecond 755nm Alexandrite Laser — Fractionated picosecond technology has been shown to lead to statistically significant improvement in atrophic, facial acne scars after 4-6 treatment sessions with minimal pain or downtime
  Other Names: Alex Laser
  Arms: Right Side Treatment with Picosecond 755NM Alexandrite laser

SUMMARY:
To assess efficacy and safety of paired picosecond 755nm Alexandrite laser with focused lens array (PSAL; Picosure®, Cynosure, Westford, MA) and radiofrequency microneedling (RFM; Potenza™, Cynosure, Westford, MA) for treatment of facial, atrophic acne scars.

DETAILED DESCRIPTION:
The primary objective of this clinical trial is to assess efficacy and safety of combination treatment with fractional picosecond 755nm Alexandrite laser with focused lens array (Picosure®, Cynosure, Westford, MA) and radiofrequency microneedling (Potenza™, Cynosure, Westford, MA) for treatment of facial, atrophic acne scarring.

Enrolled subjects will be randomized to receive picosecond 755 nm Alexandrite laser treatment to either the left or right facial half. The subjects will then undergo full face radiofrequency microneedling (RFM).

Subjects satisfying all inclusion and no exclusion criteria will be enrolled in this trial. Prior to receiving any study treatment, mandatory digital photographs will be obtained of each subject's treatment area. In order to participate in the study, subjects must provide written informed consent to have their photographs used for research, publication, and/or commercial purposes.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females aged 18 or older
* Subjects in good general health based on investigator's judgment and medical history
* Moderate to severe atrophic acne scarring on the face per ECCA (échelle d'évaluation clinique des cicatrices d'acné) acne grading scale
* Understands and accepts obligation not to receive any other procedures on the treatment area through the length of the study
* Understands and accepts the obligation and is logistically able to be present for all visits
* Is willing to comply with all requirements of the study and sign the informed consent documents
* Must be willing to maintain usual sun exposure for the duration of the study
* Subject agrees to avoid tanning or use of sunless tanner during the entire course of the study
* Negative urine pregnancy test result at the time of study entry (if applicable)
* For female subjects of childbearing potential, must be willing to use an acceptable form of birth control during the entire course of the study. All systemic birth control measures must be in consistent use for at least 30 days prior to study enrollment.

  1. A female is considered of childbearing potential unless she is postmenopausal, without a uterus and/or both ovaries, or has had a bilateral tubal ligation.
  2. Acceptable methods of birth control are: oral contraceptives, contraceptive patches/rings/implants, Implanon®, Depo-Provera®, double-barrier methods (e.g., condoms and spermicide), abstinence, and/or vasectomy of partner with a documented second acceptable method of birth control, should the subject become sexually active.

Exclusion Criteria:

* Female subjects who are pregnant, planning a pregnancy, or breast feeding during the study
* The subject is hypersensitive to light in the near infrared wavelength region
* The subject is taking medication which is known to increase sensitivity to sunlight
* The subject has a seizure disorders triggered by light
* The subject is receiving or have received gold therapy
* The subject has a pacemaker
* The subject has a metal implant that interferes with the transmission of energy to the electrical field
* The subject has any embedded electronic devices that give or receive a signal such as Implantable Cardiac Defibrillators (ICD) or Cardiac Resynchronization Therapy (CRT) devices: treatment may interfere with the functionality of the device and/or damage the electronic implant
* Gold allergy
* The subject has nerve insensitivity to heat in the treatment area or in the neutral pad placement area or a neuropathic disorder
* The subject has severe laxity or sagging that causes redundant folds of tissue or hanging skin in the area to be treated
* Dermal fillers, neuromodulator, biostimulatory injectables, fat grafting, radiofrequency device treatments, microfocused ultrasound device treatments, laser and light-based device treatments, microneedling to the face during the 6-month period before study treatment m) Subjects with tattoos in the treatment areas n) Subjects with a significant history or current evidence of a medical, psychological, or other disorder that, in the investigator's opinion, would preclude enrollment into the study
* Subjects with a history of or presence of any skin condition/disease (including but not limited to any visible rash, atopic dermatitis, psoriasis, actinic keratoses, keratinocyte carcinoma, melanoma, etc.) in the treatment area that might interfere with the diagnosis or evaluation of study parameters
* History of keloid or hypertrophic scarring
* Subjects with an active bacterial, viral, or fungal infection of the treatment areas
* The subject has a significant systemic illness, such as lupus, or an illness localized in area being treated
* History of lidocaine sensitivity deemed by the investigator to preclude the subject from enrolling into the study
* Subjects planning any cosmetic procedure to the treatment areas during the study period, other than the treatment that will be performed by the investigator
* Presence of incompletely healed wound(s) in the treatment area
* Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Volumetric analysis of change in treatment zone for acne scars using 3D imaging | Baseline, Day 7, Day 35, Day 63, Day 91, Day 121, Day 181, Day 271
  3D photography will be taken
  Standardized 3D Vectra Photography with standard lighting and camera positioning to ensure comparable before and after treatment photographs of the face. Photographs will be taken, capturing three (3) views of the hip area: anterior, right oblique (45°), and left oblique (45°). 3D photography is taken at every time frame to compare the appearance of acne scars to the previous photo.
ECCA acne grading scale by blinded investigator to assess change | Day 7, Day 35, Day 63, Day 91, Day 121, Day 181, Day 271
  Blinded Investigator ECCA (échelle d'évaluation clinique des cicatrices d'acné) acne grading scale
  V-Shaped atrophic scars, diameter of less than 2mm, and punctiform 0= no scar
  1. a few scars
  2. limited number of scars
  3. many scars
  U-shaped atropic scars, diameter of 2-4 mm, with sheer edges 0= no scar
  1. a few scars
  2. limited number of scars
  3. many scars
  M-shaped atrophic scars, diameter of more than 4mm, superficial and with irregular surface 0= no scar
  1. a few scars
  2. limited number of scars
  3. many scars
  Superficial elastolysis 0= absent
  1. mild
  2. moderate
  3. intense
  Hypertrophic inflammatory scars, scars of less than 2 years of age 0= no scar
  1. a few scars
  2. limited number of scars
  3. many scars
  Keloid scars, hypertrophic scars, of more than 2 years of age 0= no scar
  1. a few scars
  2. limited number of scars
  3. many scars
Physician Global Aesthetic Improvement Scale (PGAIS) by blinded investigator | Day 35, Day 63, Day 91, Day 121, Day 181, Day 271
  Blinded Investigator Global Aesthetic Improvement Scale Assessment (PGAIS)
  Rating Description
  1. Very Much Improved: Optimal cosmetic result in this subject.
  2. Much Improved: Marked improvement in appearance from the initial condition, but not completely optimal for this subject.
  3. Improved: Obvious improvement in appearance from initial condition, but a re-treatment is indicated.
  4. No Change: The appearance is essentially the same as the original condition.
  5. Worse: The appearance is worse than the original condition.
  Scores (write a number under each treated area or check "Not Treated") Left Facial Half Right Facial Half
  Not Treated Not Treated
Blinded Identification of correct treatment area by blinded investigator | Day 271
  The baseline (Day 0) and 6 month (Day 259) photographs will be randomly put side-by-side and labeled either (A) or (B). The blinded investigator will then fill out the following:
  1. Do you see an improvement in photoaging between the two sets of photos? (Yes / No)
  2. If yes to question #1:
     1. Which is the post-treatment photograph? (A / B)
     2. Which is the treatment side? (Right / Left)

SECONDARY OUTCOMES:
Subject Global Aesthetic Improvement Scale (SGAIS) | Day 35, Day 63, Day 91, Day 121, Day 181, Day 271
  Subject Global Aesthetic Improvement Scale Assessment (SGAIS)
  How would you rate the change in appearance of your treated areas? Non-treated areas will be checked as "Not Treated" for you.
  Rating Description
  1. Very Much Improved: Optimal cosmetic result
  2. Much Improved: Marked improvement in appearance form the initial condition, but not completely optimal
  3. Improved: Obvious improvement in appearance from initial condition
  4. No Change: The appearance is essentially the same as the original condition
  5. Worse: The appearance is worse than the original condition Scores (write a number to rate each treated area) Left Facial Half Right Facial Half
  Not Treated Not Treated
Evaluation of side effects by investigators | Day 7, Day 35, Day 63, Day 91, Day 121, Day 181, Day 271
  Treating Investigator Evaluation of Side Effects Rating Description 0 NONE: Normal
  1. TRACE: Barely visible and localized
  2. MILD: Somewhat visible and diffuse
  3. MODERATE: Visible and diffuse
  4. SEVERE: Extremely visible and dense SCORES (write number under each treated area or check "Not Treated")
  Erythema Left Facial Half Right Facial Half
  Not Treated Not Treated
  Edema Left Facial Half Left Facial Half
  Not Treated Not Treated
  Bruising/Petechiae Left Facial Half Left Facial Half
  Not Treated Not Treated
  Ulcers Left Facial Half Left Facial Half
  Not Treated Not Treated
  Hyperpigmentation/Hypopigmentation Left Facial Half Left Facial Half
  Not Treated Not Treated
Ultrasound imaging measurements of dermal edema | Day 7, Day 35, Day 63, Day 91
  Treating investigator measurement of Sub-Dermal Edema by ultrasonography
  Treating Investigator Measurement of Sub-Dermal Edema by Ultrasonography Depth of dermis (mm) Ultrasound images will be obtained at the point of intersection when a horizontal line is drawn from the ala to the tragus and a vertical line is drawn from the lateral canthus to the lateral oral commissure.
  Left Facial Half Right Facial Half

IPD SHARING:
Plan to Share IPD: Undecided